CLINICAL TRIAL: NCT06606730
Title: OPTimizing Adjuvant Prescription of PEMBROlizumab in Patients With Early-stage Triple-negative Breast Cancer Achieving Pathologic Complete Response After Standard Neoadjuvant Chemotherapy and Pembrolizumab
Brief Title: Personalizing the Use of Pembrolizumab for Patients Who Have a Strong Response in Early Triple Negative Breast Cancer
Acronym: OPT-PEMBRO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2401; 2024-515787-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancers; Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Administration of pembrolizumab for 6 months
  Interventions: Drug: Pembrolizumab
- Deescalation (Experimental): Patients will be followed up according to standard practice for 4 years
  Interventions: Other: Deescalation

INTERVENTIONS:
Drug: Pembrolizumab — Administration of pembrolizumab for 6 months
  Other Names: Keytruda
  Arms: Control
Other: Deescalation — Patients will be followed up according to standard practice for 4 years
  Arms: Deescalation

SUMMARY:
OPT-PEMBRO trial is a pragmatic, multicentre, international, prospective, non-inferiority, two-arms, randomised (1:1), open-label, Phase III clinical study.

The main goal of this research is to determine if patients with triple-negative breast cancer, who experience a complete response after neoadjuvant treatment, have the same chance of avoiding cancer recurrence whether they stop pembrolizumab or continue taking it for an additional 6 months.

This research will also take into account patients tolerance to treatment and quality of life.

DETAILED DESCRIPTION:
Triple-negative breast cancer is a particular type of breast cancer in which the cancer cells do not possess receptors for the proteins estrogen, progesterone, or HER2. The usual treatment for early-stage triple-negative breast cancer consists of chemotherapy and immunotherapy (a treatment (in this case, pembrolizumab) designed to stimulate the body's immune defenses against cancer cells) for 6 months before surgery, followed by a further 6 months of immunotherapy after surgery. Although this sequence is the reference treatment, the addition of an immunotherapy extension after surgery may not bring any additional benefit in patients who have had an excellent response to neoadjuvant treatment (before surgery), demonstrated by tumor disappearance at the time of surgery, and who therefore have a good prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent prior to any trial-related procedures. When the patient is physically unable to give his written consent, a trusted person of his choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent;
2. Age ≥ 18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
4. Histologically documented stage II-III breast cancer according to the primary tumour-regional lymph node anatomic staging criteria of the American Joint Committee on Cancer (AJCC), 8th edition as determined by the investigator during radiologic assessment, clinical assessment or both;
5. Estrogen receptor (ER) and Progesterone receptor (PR) ≤10%; HER2-negative as per ASCO/CAP guidelines Note: In case of bilateral breast cancer, participation in the study is permitted as long as both tumours are triple negative;
6. Patients previously treated with neoadjuvant chemotherapy in combination with pembrolizumab for a minimum of 6 cycles (All systemic chemotherapy must have been completed preoperatively);
7. Absence of residual invasive disease in the breast or lymph nodes after the completion of neoadjuvant therapy (Residual ductal carcinoma in situ [DCIS] is allowed);
8. Have had an adequately excised breast cancer (surgical removal of all clinically evident disease in the breast and lymph nodes) :

   1. Breast surgery: patients must have undergone either breast-conserving surgery or total mastectomy with histologically negative margins for invasive tumour and DCIS. Patients with margins positive for lobular carcinoma in situ (LCIS) are eligible without additional resection.
   2. Lymph node surgery: patients must have had sentinel lymph node biopsy (SLNB) and/or axillary lymph node dissection (ALND) to evaluate the pathologic nodal status;
9. Patients that have received adequate locoregional radiation therapy or with planned adequate locoregional radiation therapy;
10. Adequate organ and bone marrow functions. All screening lab tests should be performed within 28 days before randomisation;

    1. Absolute Neutrophil Count (ANC) ≥ 1,000 /µL
    2. Platelets ≥ 100,000 /µL
    3. Hemoglobin ≥ 9 g/dL
    4. Creatinine clearance ≥ 30 mL/min for subject with creatinine levels > 1.5 x institutional upper limit of normal (ULN)
    5. Total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN (Patients with Gilbert's disease with a total bilirubin ≤ 2.5 x ULN and direct bilirubin within normal limits are permitted)
    6. Aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤ 2.5 x ULN
11. Randomisation must take place no more than 12 weeks after breast surgery. Adjuvant radiotherapy is authorized. If given, as per investigator discretion it can be given concurrently with pembrolizumab;
12. Patients must not be pregnant or nursing (for women of childbearing potential only, a negative serum pregnancy test must be obtained within 7 days of Cycle 1 Day 1);
13. Women of childbearing potential and male patients must agree to use 1 effective form of contraception and up to 4 months after the last dose of study drugs;
14. Patients should be able and willing to comply with study visits and procedures as per protocol;
15. Patients must be affiliated to a Social Security System (or equivalent).

Exclusion Criteria:

1. Radiological or clinical evidence of metastatic disease (stage IV) documented by imaging or clinical examination;
2. Evidence of recurrent disease following preoperative therapy and surgery;
3. Any prior history of (ipsi- or contralateral) invasive breast cancer;
4. Patients with a prior or concurrent malignancy (other than invasive breast cancer) whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of the investigational regimen;
5. Patients for whom pembrolizumab has been permanently discontinued during the neoadjuvant phase of treatment due to pembrolizumab-related AE;
6. History of intolerance, including Grade 3 or 4 infusion reaction or hypersensitivity to pembrolizumab or murine proteins or any component of the product;
7. Medical conditions that require chronic systemic steroids (> 10 mg prednisone or equivalent) or any other form of immunosuppressive medication in the past 2 years. Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment;
8. Known active liver disease, e.g. due to HBV, HCV, autoimmune hepatic disorders, or sclerosing cholangitis;
9. HIV-infected patients on effective anti-retroviral therapy with detectable viral load within 6 months prior to enrollment;
10. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better;
11. Patients unwilling or unable to comply with the medical follow-up required by the trial due to geographic, familial, social, or psychological reasons;
12. Persons deprived of their liberty or under protective custody or guardianship;
13. Participation in another therapeutic trial within the 30 days prior to randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2454 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2033-01-01 (Estimated); Study Completion 2039-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | From randomization to disease progression or death, up to 8 years.
  Recurrence-free survival is defined as the time from randomisation to invasive loco-regional or distant recurrence or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Acute and late toxicity during the study | Throughout study, up to 1 year.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders
Patient reported outcome (PRO)-CTCAE composite score | At baseline, 12 weeks, end of treatment, 1 year after end of treatment, 2 years after end of treatment and 3 years after end of treatment
  The PRO-CTCAE composite score is a self-reported questionnaire to assess selected adverse events (bloating, diarrhea, abdominal pain, rash, itching, anorexia, nausea, fatigue, dyspnea, radiation skin reaction, myalgia, arthralgia, pain, and peripheral sensory neuropathy)
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 12 weeks, end of treatment, 1 year after end of treatment, 2 years after end of treatment and 3 years after end of treatment
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire - Breast cancer module (QLQ-BR42) | At baseline, 12 weeks, end of treatment, 1 year after end of treatment, 2 years after end of treatment and 3 years after end of treatment
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR42 incorporates nine multi-item scales to assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. Higher scores indicate more severe symptoms or problems for all items.
The developed 5-level version of EQ-5D (EQ-5D-5L) | At baseline, 12 weeks, end of treatment, 1 year after end of treatment, 2 years after end of treatment and 3 years after end of treatment
  Developed by the EuroQol group, the self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials consists of a descriptive system and a visual analogue scale (VAS).
  The EQ-5D-5L descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each dimension has 5 levels (1 = "no problems", 2 = "slight problems", 3 = "moderate problems", 4 = "severe problems", and 5 = "extreme problems"). This questionnaire provide a 5-digit score which generate a health state profile. The VAS records the patient's self-rated health on a vertical visual analogue scale where the score range from 0 (The best health you can image) to 100 (The worst health you can image). The VAS is used as a quantitative measure of health outcome that reflects the patient's own judgement.
Impact of Cancer Version 2 (IOC v2) Question 11 | At baseline, 12 weeks, end of treatment, 1 year after end of treatment, 2 years after end of treatment and 3 years after end of treatment
  The Impact of Cancer Version 2 (IOCv2) is a 47-item questionnaire. The question 11 is concerning fear of recurrence.
  The item is scored on a five-point scale (1 = "strongly disagree", 2 = "disagree", 3 = "neutral", 4 = "agree", and 5 = "strongly agree"). Higher scores on the positive impact indicate greater positive impacts, while higher scores on the negative impact indicate greater negative impacts.
Menstruation recovery rate | Throughout the study completion, up to 8 years.
  Menstruation recovery rate refers to how quickly or how often a patient returns to having regular menstrual periods after experiencing a disruption.
Impact on pregnancy | Throughout the study completion, up to 8 years.
  The impact of the treatment strategy on pregnancy is defined as the number of patient becoming pregnant and the outcomes (healthy birth, miscarriage, stillbirth, preterm birth, and complications) at the end of the pregnancy.
LHRH agonist prescription | Throughout the study completion, up to 8 years.
  Patterns of use of LHRH agonist during adjuvant pembrolizumab treatment.
Invasive breast cancer-free survival (IBCFS) | From randomization to IBCFS or death, up to 8 years.
  Invasive breast cancer-free survival (IBCFS) is defined as the time from randomization to invasive ipsilateral or contra-lateral breast tumour recurrence, loco-regional invasive recurrence, distant recurrence, and death from breast cancer, death from non-breast cancer or from an unknown cause.
Distant relapse free-survival (DRFS) | From randomization to distant recurrence or death, up to 8 years.
  Distant relapse free-survival (DRFS) is defined as the time from randomization to distant recurrence, death from non-breast cancer or from an unknown cause.
Incidence of second primary cancer | From randomization to apparition of a second cancer, up to 8 years.
  Incidence of second primary cancer is defined as the diagnostic of a completely different type of cancer (i.e other than breast)
Overall survival (OS) | From randomization to death, up to 8 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Cost-effectiveness analysis of the proposed therapeutic strategy (ISPOR-model) | Throughout the study completion, up to 8 years.
  The economic cost of the pembrolizumab as compared to observation will be evaluated using an International Society for Pharmacoeconomics and Outcomes Research (ISPOR) standard health economic decision model. The cost of pembrolizumab and other concomitant treatment will be analysed based on country specific guidelines together with survival data to represent the clinical pathway for early breast cancer in each country. Results will be expressed in terms of cost assessments, incremental cost-effectiveness ratio and quality of life adjusted life years.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Mourato Ribiero, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (2):
- Cliniques Universitaires Saint Luc Brussels, Brussels, Belgium
- Institut Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No